CLINICAL TRIAL: NCT05625867
Title: Post-Resuscitation Interdisciplinary Consultation System: a Randomized, Multicenter, Interventional Study to Assess Quality of Life After a Stay in the COPRéa Intensive Care Unit
Acronym: COPRéa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LAURENT UB 2022
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Post Intensive Care Syndrome
MeSH Terms: conditions — postintensive care syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Post-resuscitation interdisciplinary consultation at 4/5 months after discharge from the ICU (Experimental)
  Interventions: Other: Psychological and quality of life questionnaires; Other: Interdisciplinary consultation at 4/5 months
- Patient managed under standard practice conditions (Active Comparator)
  Interventions: Other: Psychological and quality of life questionnaires

INTERVENTIONS:
Other: Psychological and quality of life questionnaires — At 4/5 months and at 9 months
Other: Interdisciplinary consultation at 4/5 months — About ten days after the questionnaires were administered
  Arms: Post-resuscitation interdisciplinary consultation at 4/5 months after discharge from the ICU

SUMMARY:
A patient's stay in the ICU is not without consequences and can cause various physical and/or psychological sequelae such as anxiety, depression, post-traumatic stress disorder (PTSD), physical weakness and memory problems. These sequelae are grouped under the name "post intensive care syndrome" or PICS.

Numerous studies have shown that PICS affects 50-70% of patients; however, very few studies have been conducted on the medical and psychological support devices needed for these patients following their hospitalization. Despite recommendations to set up an early and specific rehabilitation program, post-resuscitation consultations are not very frequent in France. The aim of the study is to measure the impact of an interdisciplinary post-resuscitation consultation on the quality of life of patients who have stayed more than 6 days in an intensive care unit.

All patients who agreed to participate will be followed for a period of 9 months after discharge from the ICU.

One month after discharge from the ICU, the patients will be randomly assigned to

* either in the "intervention" group who will benefit from an interdisciplinary post resuscitation consultation 4/5 months after their discharge from the intensive care unit
* or in the "control" group without post resuscitation consultation. They will all be contacted at 4/5 and 9 months to complete psychological and quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Person who has given oral consent
* Patient 18 years of age or older
* Patient with at least one organ failure
* Patient with a stay of 6 days or more

Exclusion Criteria:

* Person who is not affiliated or not a beneficiary of a social security system
* Patient at the end of his/her life
* Patient who does not speak French
* Minor (< 18 years old)
* Person subject to a legal protection measure (curatorship, guardianship)
* Person subject to a legal protection measure
* Pregnant, parturient or breastfeeding women
* Patient incarcerated
* Patient with a psychiatric history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Estimated)
Dates: Start 2023-02-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
MOS SF-36 Quality of Life Scale Score | Between 4/5 and 9 months after discharge from intensive care

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No